CLINICAL TRIAL: NCT07100899
Title: Effects of Dual Task Training Versus Task-specific Training on Lower Limb Function, Trunk Control and Balance in Chronic Stroke Patients: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmed Alshimy (Other)
Responsible Party: Sponsor-Investigator, Ahmed Alshimy, Lecturer of Physical Therapy for Neurology and it's Surgery, AlRyada University for Science & Technology
Organization: AlRyada University for Science & Technology (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/ 012/003564
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Stroke
Keywords: Stroke; dual task training; task-specific training; lower extremity; balance; trunk control
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): received dual motor task training in addition to the selected physiotherapy program, three times a week for twelve weeks, with each session lasting sixty minutes.
  Interventions: Other: Dual task training; Other: Selected physiotherapy program
- Group B (Experimental): received task-oriented training in addition to the selected physiotherapy program, three times a week for twelve weeks, with each session lasting sixty minutes.
  Interventions: Other: Task-specific training; Other: Selected physiotherapy program
- Group C (Other): only received the selected physiotherapy program, three times a week for twelve weeks, with each session lasting sixty minutes.
  Interventions: Other: Selected physiotherapy program

INTERVENTIONS:
Other: Dual task training — Dual motor task training for 30 minutes. The dual motor training was divided into two phases. The first part involved a single task condition in which the stroke patient was instructed to stand up from a seated position at a self-selected speed without the use of upper limb assistance. Cognitive and physical tasks, is the second part of training. In addition to a 30-minute selected physiotherapy program.
  Arms: Group A
Other: Task-specific training — Began with a highchair before switching to a low one. In addition to a 30-minute selected physiotherapy program.
  Arms: Group B
Other: Selected physiotherapy program — Consisting of trunk control, trunk stabilization, balance training and lower extremity strengthening exercises (primarily for the hip adductors and abductors) for 60 minutes.

SUMMARY:
One of the leading causes of disability among the elderly is stroke. After a stroke, it is highly usual for lower extremity function, balance and trunk control to be compromised. After a stroke, trunk control is a crucial early predictor of functional recovery. Following a stroke, proximal trunk control is necessary for distal limb movement control, balance, and functional capacity.

DETAILED DESCRIPTION:
Forty-five chronic stroke patients, ages 45 to 55, were divided into three equal groups for this randomized controlled study: GA consisted of 15 patients, GB of 15 patients, and GC of 15 patients each. Group A (the study group) received dual motor task training in addition to the selected physiotherapy program, Group B (the study group) received task-oriented training in addition to the selected physiotherapy program, and Group C only received the selected physiotherapy program for 12 weeks. All groups received treatment three times a week for twelve weeks, with each session lasting sixty minutes. The Trunk Impairment Scale (TIS), Functional Reach Test (FRT), Biodex Balance System (BBS), and Fugl Meyer Lower Extremity (FM-LE) were used to evaluate each of the three groups pre and post treatments.

ELIGIBILITY:
Inclusion Criteria:

* 45 chronic stroke patients between the ages of 45 and 55 who were of both sexes, had been ill with stroke for more than six months to a year, had received at least nine years of education, had a score on the Berg balance scale between 41 and less than 45, and had cognitive functions greater than 26 on the MOCA scale were included in this study

Exclusion Criteria:

* Patients who had any neurological condition that affected balance other than stroke (such as inner ear, vestibular, or cerebellar dysfunction), communication disorders, uncontrolled hypertension, diabetes, or unstable angina, hearing or vision issues, or respiratory disorders were not allowed to participate.

Ages: 45 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2025-06-05 (Actual); Primary Completion 2025-07-05 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
Trunk impairment scale | 4 weeks
  It assesses trunk coordination skills as well as static and dynamic balance while seated
Functional Reach test | 4 weeks
  This one-item exam is intended to serve as a rapid screening tool for balance issues
Biodex Balance System | 4 weeks
  Used to evaluate balance
Fugl-Meyer lower extremity | 4 weeks
  This test is designed to evaluate lower extremity motor and sensory impairment after a stroke

CONTACTS AND LOCATIONS:
Locations (1):
- Al Ryada University for Science and Technology, Sadat, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: No